CLINICAL TRIAL: NCT00275938
Title: A Pilot Study Of Interferon Alpha 2b Plus Ribavirin In The Treatment Of Patients With Chronic Hepatitis B
Brief Title: Interferon Alpha 2b Plus Ribavirin for Chronic Hepatitis B
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Schering-Plough (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 145R3
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Last update posted 2006-01-12 (Estimated); Status verified 2006-01

CONDITIONS: Chronic Hepatitis B
Keywords: hepatitis B virus; e antigen; interferon; ribavirin
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — Interferon alpha-2; Ribavirin

INTERVENTIONS:
Drug: interferon alpha 2b plus ribavirin
Drug: interferon alpha 2b plus placebo

SUMMARY:
Hepatitis B virus (HBV) causes a wide spectrum of liver diseases, such as fulminant or acute hepatitis, chronic hepatitis, liver cirrhosis, and hepatocellular carcinoma. The number of individuals infected with this virus has been estimated to be as high as 350 million. Thus, in addition to global hepatitis B vaccination, effective treatment of chronic hepatitis B is also needed.

Currently, there are no effective antiviral treatments to cure HBV infection in patients with chronic hepatitis B. Five drugs have been approved for the treatment of chronic hepatitis B at present: conventional interferon (IFN) alpha, lamivudine, adefovir dipivoxil, pegylated IFN alpha and recently entecavir. Overall, satisfactory virologic and serologic responses could be achieved using pegylated IFN alpha alone in around 20-44% of these patients. Nevertheless, better treatment options are still needed for the remaining >50% non-responders.

Although the best treatment choice for chronic hepatitis B is not clarified yet, certain therapeutic concepts could be derived from the experience of treating patients with chronic hepatitis C. A major advancement in treating hepatitis C virus (HCV) infection has been the development of combination therapy with IFN and ribavirin. IFN monotherapy is limited by poor sustained virologic responses, even when higher doses of IFN are used. IFN plus ribavirin combination therapy, in contrast, results in much improved treatment outcomes. In our previous study and others, sustained remission rate after cessation of therapy were significantly higher in patients receiving combination therapy than those receiving IFN alone. Therefore, combination therapy with IFN and ribavirin has been recommended as the standard treatment regimen for chronic hepatitis C. Furthermore, we have used ribavirin and IFN combination for the treatment of dual chronic hepatitis B and C, and the results also revealed that the efficacy of clearing HCV RNA was not affected by the presence of HBV infection. Interestingly, after a little more than 2-year post-treatment follow-up, we found that a significant portion (21%) of the responsive patients also cleared HBsAg. These findings imply that this combination regimen might be also effective for the control of chronic hepatitis B. We thus conducted a randomized, multi-center, placebo-controlled study in patients with HBeAg-positive chronic hepatitis B.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) causes a wide spectrum of liver diseases, such as fulminant or acute hepatitis, chronic hepatitis, liver cirrhosis, and hepatocellular carcinoma. The number of individuals infected with this virus has been estimated to be as high as 350 million. Thus, in addition to global hepatitis B vaccination, effective treatment of chronic hepatitis B is also needed.

Currently, there are no effective antiviral treatments to cure HBV infection in patients with chronic hepatitis B. Five drugs have been approved for the treatment of chronic hepatitis B at present: conventional interferon (IFN) alpha, lamivudine, adefovir dipivoxil, pegylated IFN alpha and recently entecavir. Conventional IFN alpha monotherapy has a narrow range of efficacy. Lamivudine, is relatively cheaper, better tolerated, and has been shown to be effective in patients with both hepatitis B e antigen (HBeAg)-positive and -negative chronic hepatitis B. However, virologic response to lamivudine is not as durable as that occurred spontaneously or induced by IFN treatment. In addition, prolonged lamivudine treatment is commonly associated with the emergence of drug-resistance HBV mutants accompanied by the development of breakthrough hepatitis. Adefovir is potent and has been approved for the treatment of chronic hepatitis B in several countries, but is nephrotoxic at daily doses higher than 10 mg and is still not available widely. Entecavir, a carbocyclic deoxyguanosine analog, which is active against both lamivudine- and adefovir dipivoxil-resistant HBV, is the most potent anti-HBV agent ever discovered,11 however, its long-term efficacy remains to be evaluated. Pegylated IFN alpha has recently been shown to be superior to conventional IFN alpha and lamivudine, and has also been approved for the treatment of chronic hepatitis B. Overall, satisfactory virologic and serologic responses could be achieved using pegylated IFN alpha alone in around 30-44% of these patients. Nevertheless, better treatment options are still needed for the remaining >50% non-responders.

Although the best treatment choice for chronic hepatitis B is not clarified yet, certain therapeutic concepts could be derived from the experience of treating patients with chronic hepatitis C. A major advancement in treating hepatitis C virus (HCV) infection has been the development of combination therapy with IFN and ribavirin. IFN monotherapy is limited by poor sustained virologic responses, even when higher doses of IFN are used. IFN plus ribavirin combination therapy, in contrast, results in much improved treatment outcomes. In our previous study and others, sustained remission rate after cessation of therapy were significantly higher in patients receiving combination therapy than those receiving IFN alone. Therefore, combination therapy with IFN and ribavirin has been recommended as the standard treatment regimen for chronic hepatitis C. Furthermore, we have used ribavirin and IFN combination for the treatment of dual chronic hepatitis B and C, and the results also revealed that the efficacy of clearing HCV RNA was not affected by the presence of HBV infection. Interestingly, after a little more than 2-year post-treatment follow-up, we found that a significant portion (21%) of the responsive patients also cleared HBsAg. These findings imply that this combination regimen might be also effective for the control of chronic hepatitis B. We thus conducted a randomized, multi-center, placebo-controlled study in patients with HBeAg-positive chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female, 18 to 60 years of age chronic hepatitis B patients Patient must have documented positive serum HBsAg for a minimum of 6 months prior to entry into study.

Patients must show evidence of HBV replication and hepatitis documented by Positive serum HBV-DNA within 3 months prior to entry (HBV-DNA > 2.5 pg/ml) Positive serum HBeAg within 3 months prior to entry. Documented presence of abnormal alanine aminotransferase (ALT) twice within 3 months prior to entry (2 to 10 fold above the upper normal level) Liver biopsy finding shows chronic hepatitis without liver cirrhosis

Compensated liver disease with the following minimum hematological and serum biochemical criteria:

* Hemoglobin values of ≥ 12 gm/dL for both sexes
* WBC ≥ 3,000/mm3
* Neutrophil count ≥ 1,500/ mm3
* Platelets ≥ 100,000/ mm3
* Total bilirubin ≤ 2 mg/dL
* Albumin ≥ 3.5 g/dL
* Uric acid within normal ranges
* Serum creatinine ≤ 123.76 mmol/L (≤1.4 mg/dL)
* Fasting blood sugar ≤ 6.38 mmol/L (≤115 mg/dL) for non-diabetic patients
* Hemoglobin ≤ 8.5% for diabetic patients (whether on medication and/or controlled with diet) Thyroid Stimulating Hormone (TSH), T3 & T4 within normal limits Negative serum antibody to hepatitis C Negative antibody to human immunodeficiency virus (anti-HIV) ELISA method If the patient has a history of diabetes or hypertension, a baseline ocular examination will be required.

Alfa-fetoprotein within normal range Written informed consent



Exclusion Criteria:

* Patients older than 60 years of age

Any cause for the liver disease based on patient history or biopsy (where applicable) other than chronic hepatitis B, including but not limited to:

Co-infection with HCV and/or HIV Hemochromatosis (iron despistion > 2 + in liver parenchyma) Alpha-1 antitrypsin deficiency Wilson's disease Renal or liver transplant patients Autoimmune hepatitis Alcoholic liver disease Obesity related liver disease Drug related liver disease Evidence of decompensated liver disease such as history or presence of ascites, bleeding varices, hepatic encephalopathy.

Any known pre-existing medical condition that could interfere with the patient's participation in and completion of the treatment such as:

Pre-existing psychiatric condition, especially severe epression, or a history of severe psychiatric disorder CNS trauma or active seizure disorders requiring medication. Patients with any history of cardiovascular dysfunction. Patients with any hemoglobinopathy including but not limited to thalassemia major and minor Poorly controlled diabetes mellitus Chronic pulmonary disease Immunologically mediated disease Clinical gout Sexually active females of childbearing potential must be practicing adequate contraception, Sexually active males must be practicing acceptable methods of contraception (vasectomy, condom + spermicide, monogamous relationship with a female partner who practices an acceptable method of contraception) during the treatment period and for 6 months after discontinuation of therapy.

Female patients must not breast feed during the treatment period. Patients must agree to limit the drinking of alcohol during the course or the treatment.

Patients receiving Chinese herbal medication during the past 3 months prior to study entry.

Patient who did not respond to previous interferon therapy or who relapsed after a previous course of Interferon therapy.

Patients who have been enrolled in any clinical trial for the treatment of chronic hepatitis B.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120
Dates: Start 1998-10; Study Completion 2001-06

PRIMARY OUTCOMES:
Undetected serum HBV DNA level (i.e. less than 2.5 pg/ml) at the end of the 24-week follow-up period

SECONDARY OUTCOMES:
HBV DNA level at the end of treatment
clearance of HBeAg and rate of ALT normalization both at the end of the 32-week treatment period and at the end of the 24-week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yang Lai, Professor, Principal Investigator — National Taiwan University Hospital